CLINICAL TRIAL: NCT00786045
Title: Fitness Intervention Tiral for Stroke: Enhancing Walking Endurance Using Home Rehabilitation Programs
Brief Title: Fitness Intervention Trial for Stroke
Acronym: FITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Nancy Mayo, BSc(PT), MSc, PhD, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: A11-M107-02A; MCT_66794
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; walking
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home Cycling Program (Experimental): Participants will be given a time and intensity graded program at an intensity that is comfortable and tolerable for the individual. The individual will be encouraged to augment, gradually, either the time of cycling per day or the work of cycling, always keeping within the limits of comfort and tolerability. Participants will also be given a target heart rate threshold to try and meet but not to exceed. This will be based their response to the stress test and will most likely be between 50% and 70% of maximum age-predicted heart rate. The aim is to build up to one-half hour of cycling per day. All bicycles will be equipped with electronic monitoring of speed, distance, and heart rate.
  Interventions: Other: Home Cycling Program
- Control (No Intervention): The investigators have devised a series of mobility-related tasks that can be easily and safely carried out at home without ongoing professional supervision

INTERVENTIONS:
Other: Home Cycling Program — Participants will be given a time and intensity graded program at an intensity that is comfortable and tolerable for the individual. The individual will be encouraged to augment, gradually, either the time of cycling per day or the work of cycling, always keeping within the limits of comfort and tolerability. Participants will also be given a target heart rate threshold to try and meet but not to exceed. This will be based their response to the stress test and will most likely be between 50% and 70% of maximum age-predicted heart rate. The aim is to build up to one-half hour of cycling per day. All bicycles will be equipped with electronic monitoring of speed, distance, and heart rate.
  Arms: Home Cycling Program

SUMMARY:
The objective of this study is to evaluate, among persons who have completed the restorative phase of stroke and have ceased rehabilitation, the relative effectiveness in improving functional exercise capacity of two programs for continued care, a home-based general fitness training program using stationary cycling and a disability targeted, home-based exercise program to enhance mobility and walking competency. capacity compared with the "walking" group and that consequently the cycle group will achieve a higher quality of life.

A secondary objective is to explore factors associated with compliance with the exercise regimens. Previous research has indicated that cognitive-affective-behavioural profile is related to exercise activity in a number of populations including sedentary adults, older adults and patients with cardiovascular disease. As we anticipate that one of the mechanisms by which the cycling will result in an outcome better than the more traditional type of disability tailored exercise program is through greater compliance, this second objective is very relevant. This study will also address the impact of regular exercise on cardio-vascular risk factor profile.

DETAILED DESCRIPTION:
The specific clinical hypothesis to be tested is that, over a one year period, persons assigned to the general fitness "cycle" group will experience a greater increase in functional exercise

ELIGIBILITY:
Inclusion Criteria:

* verified stroke requiring hospital admission (based on clinical and radiological evidence)
* ability to walk a minimum of 10 meters independently, using an aid or orthotic, with or without supervision,
* less than one year since the last cerebrovascular event at the time of recruitment,
* discharge from active rehabilitation (usually around 3 to 4 months post-stroke but not less than 1 month) into the geographic study area of greater Montreal and greater Halifax.

Exclusion Criteria:

* severe cognitive deficits as evaluated by the Telephone Version of the Mini-Mental State Examination such that the subject does not understand their participation in the study,
* receptive aphasia as evaluated by the Canadian Neurological Scale48 or the treating speech therapist,
* illness or disability precluding participation in either rehabilitation intervention.
* failure to pass a standard cardiology orientated history and physical examination complemented by a baseline screening exercise stress test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Functional Walking Capacity (6 Minute (walk test) | baseline, 1 month, 6 months, 12 months

SECONDARY OUTCOMES:
Quality of Life (SF-36) | Baseline, 1 month, 6 month, 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Mayo, PhD, Principal Investigator — McGill University, Division of Clinical Epidemiology
Locations (1):
- McGill University-Royal Victoria Hospital Site, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Mayo NE, MacKay-Lyons MJ, Scott SC, Moriello C, Brophy J. A randomized trial of two home-based exercise programmes to improve functional walking post-stroke. Clin Rehabil. 2013 Jul;27(7):659-71. doi: 10.1177/0269215513476312. Epub 2013 Mar 15. PMID 23503738